CLINICAL TRIAL: NCT06078618
Title: Place of Birth and Neonatal Health in Cases of Preterm Birth Between 32 and 36 Weeks of Amenorrhoea: a National Population-based Study
Brief Title: Place of Birth and Neonatal Health in Cases of Premature Birth Between 32 and 36 Weeks of Amenorrhoea
Acronym: PREM3236
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DESPLANCHES APJ 2021
Record Dates: First submitted 2023-10-03; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Premature Between 32 and 36 Weeks of Amenorrhoea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort: Mothers and their newborn babies (live or stillborn) who were delivered between 32 and 36 weeks' gestation

SUMMARY:
Moderate and late premature babies (32-36 weeks of amenorrhoea) account for around 6% of births, but 20% of neonatal deaths. These children also have an increased risk of neonatal morbidity and long-term neurodevelopmental sequelae compared with full-term newborns.

In the case of preterm birth, optimal antenatal, birth and postnatal management is necessary to prevent neonatal complications and mitigate longer-term consequences. However, we lack knowledge about the management of this at-risk population and the factors influencing their health.

This knowledge is needed in the current context of unfavourable trends in neonatal health. Over the last ten years, neonatal and infant mortality has stagnated in France, with France falling behind other European countries. According to the latest European report, France ranks 22nd out of 33 countries. The causes of this stagnation are not well known, but many hypotheses have been put forward, including sub-optimal organisation of care.

ELIGIBILITY:
Inclusion Criteria:

* All mothers and their newborn babies (live or stillborn) who had a delivery stay between 32 and 36 days of age recorded in the PMSI between 01/01/2015 and 31/12/2020.

Exclusion Criteria:

* Births in very small maternity units
* Births in hospitals without an obstetrics unit
* Births outside hospitals.

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective cohort based on an extraction from the National Health Data System (SNDS) and including all pregnant women giving birth between 32 and 36 completed weeks of amenorrhoea, between 1st January 2015 and 31st December 2020 in France and their newborn babies (live or stillborn).
Sampling Method: Non-Probability Sample
Enrollment: 240000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate | up to 28 days after birth
  Mortality (stillbirths, neonatal mortality before 28 days, hospital mortality)
Neonatal morbidity rate | up to 28 days after birth
  Neonatal morbidity. Composite indicator of neonatal morbidity defined by 18 ICD 10 and/or CCAM diagnostic codes and including the following sub-categories: respiratory, infectious, neurological, metabolic pathologies and obstetric trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France